CLINICAL TRIAL: NCT03706131
Title: The Effect of Cervical Mobilization on Balance and Spasticity in Multiple Sclerosis Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, ECEM KARANFİL, Research Assistant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: KA-17087
Record Dates: First submitted 2018-08-09; First posted 2018-10-15 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Multiple Sclerosis; Balance; Distorted
Keywords: multiple sclerosis; cervical region; balance; spasticity; mobilisation
MeSH Terms: conditions — Multiple Sclerosis; Muscle Spasticity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Spasticity evaluations will be done by blind investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): one session 15 minutes cervical mobilisation and home exercise
  Interventions: Other: cervical mobilisation
- control grup (No Intervention): no intervention

INTERVENTIONS:
Other: cervical mobilisation — manual therapy
  Arms: experimental group

SUMMARY:
Taking into consideration the effects of mobilization on muscle tone and balance, it is predicted that this method will have effective results in the treatment of individuals with MS. Therefore, it is thought that grade A and grade B mobilization applications can be used to strengthen the balance control mechanisms of MS individuals and to regulate muscle tone by increasing the proprioceptive input. In this study, it was aimed to investigate the short-term effects of cervical mobilization on balance and spasticity in MS individuals.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a chronic, inflammatory, demyelinating, and neurodegenerative disease of the central nervous system (CNS). The etiology of the disease is not fully known. It is thought that both autoimmune and neurodegenerative mechanisms can play a role in MS. Genetic and environmental factors are also influenced by the emergence of the disease. Although the factors that trigger MS are not fully known, autoreactive T cells and antibodies against SSS are thought to have a major pathogenic role in the development of inflammation and tissue damage. The same mechanism is held responsible for the progression of neurological disorders and functional deficits.

MS can severely limit the quality of life in patients due to the accumulation of sequelae following the attacks or the development of a progressive degenerative process, leading to progressive disability.

The disease has marked clinical heterogeneity. This difference may be in the age of onset, onset, frequency, severity and sequelae of exacerbations, worsening prevalence and cumulative impairment over time. Although there are differences in clinical and pathologic findings, variable clinical features reflect multifocal SSS destruction. In patients, somatosensory findings (burning, numbness, tingling, deep and superficial sensory deficits), motor findings (spasticity due to corticospinal involvement, muscle strength losses), postural control and coordination disorders, bladder-bowel problems, visual, cognitive and psychiatric manifestations, fatigue and sleep disorders.

Spasticity is one of the most common physical disorders in MS. It is known that 60-90% of individuals with MS develop spasticity. MS-associated spasticity; generalized, focal (which affects a part of the extremity) or multifocal (which affects more than one part of the extremities or extremities). Spasticity; due to force imbalance between agonist and antagonist muscles, affecting static joint positions and dynamic limb movements, resulting in abnormal postural conditions and stiffness. Spasticity is directly related to disease progression and muscle weakness leads to secondary fatigue due to increased energy expenditure. Depending on the spasticity, structural changes of muscles, tendons and joints affect the movements and functions of the extremities.

Equilibrium losses are one of the other important symptoms seen in MS patients, affecting about 75% of patients. Balance; the ability to keep the center of gravity of the body within the limits of the support surface. The sensory components of the balance; visual, vestibular and somatosensory system information. The feeling of proprioception, which is part of the somatosensory system; joints and extremities, which are formed by receptors located in the joints and tissues and provided by neural inputs. Proprioceptors are specific receptors that are located at different rates in different structures and tissues of the body. It is known that the cervical region is very rich in these receptors. In this respect, the neck plays a very important role in maintaining the right orientation, balance, and accordingly motor coordination of the whole body. For example; In the impaired proprioceptive processes of the lower extremities, compensation is provided by proprioceptive inputs from the cervical region to maintain body balance. The cervical region is closely related to the vestibular system, which is another sensory component of balance. This relationship is extremely important in the activity of cervico-colic (CCR) and vestibulo-colic reflexes (VCR). VCR is semicircular canal and macular origin. They are effective on the receptors on the inner ear and on the muscular extensor muscles. In one study, when vestibular stimulation accompanied the tension of the neck muscles, the sagittal VCR in the semispinalis capitis muscle increased about three-fold normally. Strengthening of the VCR reflex with tongue proprioceptive afferents is the result of summing up of CCR and VCR induced by stretching of the neck muscles. The interaction between the two reflexes showed that not only the vestibular stimulation but also the length of the neck muscles were important in the normal movement of the head over the neck.

In the treatment of spasticity and balance disorders, which are very common and difficult to manage in MS patients, drug therapies, botulinum toxin treatments, surgical treatments and physiotherapy and rehabilitation approaches are included.Physiotherapy applications; sensory, walking parameters, extremity functions, muscle tone, body and standing balance are known to have positive effects. The use of somatosensory strategies, balance exercises, coordination training, spinal stabilization exercises and activity based exercises are the physiotherapy approaches used in balance training. Mobilization techniques, which are another physiotherapy application, restoration of joint motion with the application of different forms of active and passive exercise. Mobilization is a repetitive passive motion within the limits of normal joint motion, without exceeding this limit, at different amplitudes at low speeds. The neurophysiological effects of mobilization are to improve the proprioception sensation by stimulating receptor nerve endings in different periarticular structures, changing the range of motion, pain, muscle tone, motor control and spinal stability. Inserted stretching and pushing stimulates Type III joint receptors and golgi tendon organs. In this case relaxation occurs with temporary inhibition in the muscles. This causes an increase in joint motion and prepares the joint for more stretching and mobilization. Thus, pain and protective muscle spasm are reduced. Neurophysiological effects of mobilization; decreased pain and muscle tone, postural control and balance effects.

Mobilization techniques are classified into 3 groups according to severity and degree. These; grade A (mobilization), grade B (mobilization) and grade C (manipulation). Grade (mobility); active, or active assisted movements within painless range of motion. Grade B (mobility); is a special continuous stretching technique which causes the prolongation of the connector touch. At the spinal joints, the joint is applied at the end of the range of motion. Grade C (manipulation); passive movement in the form of a minimal amplitude, high velocity push applied between the physiological boundary and the anatomical boundary.

Taking into consideration the effects of mobilization on muscle tone and balance, it is predicted that this method will have effective results in the treatment of individuals with MS. Therefore, it is thought that grade A and grade B mobilization applications can be used to strengthen the balance control mechanisms of MS individuals and to regulate muscle tone by increasing the proprioceptive input. In this study, it was aimed to investigate the short-term effects of cervical mobilization on balance and spasticity in MS individuals.

ELIGIBILITY:
Inclusion Criteria: Between the ages of 18-65

* Expanded Disability Status Scale (EDSS) score between 2-5,
* The EDSS Cerebellar System Subscale has a Functional System Score of ˃0,
* At least one of the hip extender, Gastro-soleus and Quadriceps Femoris muscles has a spasticity of ≤2 according to the Modifiye Ashworth scale (MAS)
* If the medical condition is stable and there is no drug change in the last month,
* Vertebro-bacillus test is negative,
* have no other orthopedic problems to prevent further neurological distress and participation in the study,
* At least 24 points from the Mini Mental Test,
* They are designated as volunteers to participate in the study. -

Exclusion Criteria:

* Under age 18 and older than 65 years
* The Expanded Disability Status Scale (EDSS) score is less than 2, higher than 5,
* The EDSS Cerebellar System Subscale has a Functional System Score of 0,
* The spasticity values of the hip extender, Gastro-soleus and Quadriceps Femoris muscles are ˃2 according to the Modifiye Ashworth scale (MAS)
* The cognitive problem is that the Mini Mental Test score is below 24,
* The existence of cardiovascular, orthopedic, psychological and other problems that may prevent the completion of the assessments,
* Vertebro-bacillus test is positive,
* plaque presence of cervical and thoracal region demyelination,
* Having had an attack within the last 3 months,
* Botulinum toxin administration in the last 6 months,
* Has been admitted to the physiotherapy program in the last six months -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Computerized Dynamic Posturography | 30 minutes
  balance assessment

SECONDARY OUTCOMES:
Berg Balance Scale | 7 minutes
  The BBS is a 14-item scale that was designed to measure balance in the elderly population in a clinical setting. It has also been used to assess postural balance in people with a history of stroke and traumatic brain injury. The BBS consists of 14 different tests examining individuals' ability to sit, stand, reach, maintain single-leg stance, and turn. It rates performance on a scale from 0 (cannot perform task) to 4 (normal performance on task). In the elderly population, it has been found to be a good predictor of falling, with good validity and reliability.The total possible score ranges from 0 to 56; a score of 45 or below indicates an increased risk of falling.
Range of Motion | 10 minutes
  Goniometric measurements are used by physical therapists to quantify baseline limitations of motion, decide on appro- priate therapeutic interventions, and document the effectiveness of these interventions. This assessment is used for spasticity evaluation.
Modified Ashworth Scale | 10 minutes
  The Modified Ashworth Scale (MAS) measures resistance during passive soft-tissue stretching. It is a quick and easy measure that can help assess the efficacy of treatment.
  Scoring 0 = Normal tone, no increase in tone 1 = Slight increase in muscle tone, manifested by a catch and release or minimal resistance at the end of the range of motion (ROM) when the affected part(s) is moved in flexion or extension
  1+ = Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM 2= More marked increase in muscle tone through most of the ROM, but affected part(s) easily moved 3= Considerable increase in muscle tone, passive movement difficult 4=Affected part(s) rigid in flexion or extension.

CONTACTS AND LOCATIONS:
Overall Officials: Kadriye armutlu, prof.dr., Study Director — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Karlberg M, Magnusson M, Malmstrom EM, Melander A, Moritz U. Postural and symptomatic improvement after physiotherapy in patients with dizziness of suspected cervical origin. Arch Phys Med Rehabil. 1996 Sep;77(9):874-82. doi: 10.1016/s0003-9993(96)90273-7. PMID 8822677
- See also: pubmed — https://doi.org/10.1016/S0003-9993(96)90273-7